CLINICAL TRIAL: NCT04238715
Title: A Multicenter, Open-Label, Phase 2 Trial of E7090 in Subjects With Unresectable Advanced or Metastatic Cholangiocarcinoma With FGFR 2 Gene Fusion
Brief Title: A Study of E7090 in Participants With Unresectable Advanced or Metastatic Cholangiocarcinoma With Fibroblast Growth Factor Receptor (FGFR) 2 Gene Fusion
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7090-J000-201
Record Dates: First submitted 2020-01-22; First posted 2020-01-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cholangiocarcinoma
Keywords: E7090; Cholangiocarcinoma; Unresectable cholangiocarcinoma; Metastatic cholangiocarcinoma; Fibroblast Growth Factor Receptor 2 (FGFR2); FGFR2 gene fusion
MeSH Terms: conditions — Cholangiocarcinoma; Acrocephalosyndactylia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E7090 140 mg (Experimental): Participants will receive E7090 140 mg (milligram), tablets orally once daily (QD), in 28-days treatment cycle until disease progression, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination.
  Interventions: Drug: E7090

INTERVENTIONS:
Drug: E7090 — E7090 tablets orally.

SUMMARY:
The primary purpose of the study is to assess the objective response rate (ORR) of E7090 by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 based on independent imaging review (IIR) in participants with unresectable cholangiocarcinoma with FGFR2 gene fusion who failed gemcitabine-based combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a histologically or cytologically diagnosis of intrahepatic or perihilar cholangiocarcinoma who agree to provide archival tumor sample or residual biopsy sample, or agree with tumor biopsy.
2. Participants who have confirmed FGFR2 gene fusion of tumor by fluorescence in situ hybridization (FISH) in central laboratory. FGFR2 gene fusion confirmed by the same FISH assay in another test/study will be discussed with the sponsor and agreed on a case by case basis.
3. Participants with surgically unresectable or advanced/metastatic disease who have received at least one prior chemotherapy including gemcitabine-based combination chemotherapy (example: gemcitabine and cisplatin)

   a. Prior adjuvant chemotherapy is allowed if relapse was within 6 months after last administration.
4. Measurable disease meeting the following criteria:

   1. At least 1 lesion of >=1.0 centimeter (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI).
   2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
5. Corrected serum calcium less than or equal to (<=) upper limit of normal (ULN).
6. Phosphate <=ULN.
7. Participants with Performance Status (PS) score of 0-1 established by Eastern Cooperative Oncology Group (ECOG).
8. Participants who are expected to survive for 3 months or longer after starting administration of the investigational drug.
9. Washout period required from the end of prior treatment to the start of E7090 administration will be as follows

   1. Antibody and other investigational drugs : >=4 weeks
   2. Prior chemotherapy (except small-molecule targeted therapy), surgical therapy, radiation therapy：>=3 weeks
   3. Endocrine therapy, immunotherapy, small-molecule targeted therapy: >=2 weeks

Exclusion Criteria:

1. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example: radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
2. Concomitant active infection requiring systemic treatment (except hepatitis B or C virus-infected participants who are under anti-viral treatment).
3. Participants who test positive for human immunodeficiency virus (HIV antibody) at Screening 2.
4. Child-Pugh score B or C.
5. Moderate or severe ascites extending from the pelvis to the liver surface.
6. Following ocular disorders

   1. Current evidence of Grade 2 or higher corneal disorder
   2. Current evidence of active macula disorder (example: age-related macular degeneration, central serous chorioretinal disease)
7. Participants whose toxicity of previous treatment has not recovered to Grade 1 or lower per Common Terminology Criteria for Adverse Events (CTCAE v4.03), except for alopecia, infertility and the adverse events listed in inclusion criteria.
8. Participants with prior therapy targeting FGFR2.
9. Participants who need the use of drugs or foods that strongly inhibits or induces the metabolizing enzyme cytochrome P450 (CYP) 3A4 during study treatment (there must be a time interval of >= 7 days since the final use of these drugs or foods by the start of study treatment).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
ORR | From first dose of study drug until disease progression, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years 2 months)
  The ORR will be assessed by IIR based on RECIST version 1.1. ORR is defined as a percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). CR: disappearance of all (targeted and non-target [NT]) lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to (>=) 30 percent (%) decrease in sum of diameters of target lesions taking as reference baseline, associated to non-progressive disease (non-PD) response for (NT) lesions.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the date of first dose to the date of first documentation of disease progression or date of death from any cause, whichever occurs first (up to approximately 6 years 2 months)
  PFS will be assessed by IIR based on RECIST version 1.1. PFS is defined as the time from the date of first dose to the date of first documentation of progressive disease (PD) or date of death from any cause, whichever occurs first. PD per RECIST 1.1 is defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Duration of Response (DOR) | From the date of first documentation of CR or PR to the date of first documentation of disease progression or date of death from any cause, whichever occurs first (up to approximately 6 years 2 months)
  DOR will be assessed by IIR based on RECIST version 1.1. DOR is defined as the time from the date of first documentation of CR or PR to the date of first documentation of disease progression or date of death from any cause, whichever occurs first. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Time to Response (TTR) | from the date of first study dose to the date of first documentation of CR or PR (up to approximately 6 years 2 months)
  TTR will be assessed by IIR based on RECIST version 1.1. TTR is defined as the time from the date of first study dose to the date of first documentation of CR or PR. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Overall Survival (OS) | From the date of first dose to the date of death from any cause (up to approximately 6 years 2 months)
  OS is defined as the time from the date of first dose to the date of death from any cause. For the participants who are alive or unknown, OS is censored as the date of last known alive date.
Disease Control Rate (DCR) | From first dose of study drug until disease progression, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years 2 months)
  DCR will be assessed by IIR based on RECIST version 1.1. DCR is defined as a percentage of participants with BOR of CR, PR or stable disease (SD). The BOR of SD has to be observed greater than or equal to (>=) 7 weeks from the date of first study dose. CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.
Clinical Benefit Rate (CBR) | From first dose of study drug until disease progression, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years 2 months)
  CBR will be assessed by IIR based on RECIST version 1.1. CBR is defined as a percentage of participants with BOR of CR, PR or durable SD (dSD) (duration of SD >=23 weeks). CR: disappearance of all lesions. PR: For PR, longest diameter will be used for non-lymph target lesions but short axis is measured for lymph lesions. PR: greater than or equal to >=30% decrease in sum of diameters of target lesions taking as reference baseline, associated to non-PD response for NT lesions.

CONTACTS AND LOCATIONS:
Locations (56):
- China (32):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tsinghua Chang Gung Memorial Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijng Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical University Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen Univeristy, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Affilicataed Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan provincial people's hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow, Suzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
- Japan (24):
  - Eisai Trial Site 10, Nagoya, Aichi-ken
  - Eisai Trial Site 16, Kashiwa, Chiba
  - Eisai Trial Site 11, Matsuyama, Ehime
  - Eisai Trial Site 14, Matsuyama, Ehime
  - Eisai Trial Site 2, Sapporo, Hokkaido
  - Eisai Trial Site 8, Kanazawa, Ishikawa-ken
  - Eisai Trial Site 7, Yokohama, Kanagawa
  - Eisai Trial Site 23, Tsu, Mie-ken
  - Eisai Trial Site 22, Sendai, Miyagi
  - Eisai Trial Site 13, Hirakata, Osaka
  - Eisai Trial Site 17, Suita, Osaka
  - Eisai Trial Site 9, Sunto-gun, Shizuoka
  - Eisai Trial Site 5, Bunkyo-ku, Tokyo
  - Eisai Trial Site 4, Chuo-ku, Tokyo
  - Eisai Trial Site 6, Koto-ku, Tokyo
  - Eisai Trial Site 3, Mitaka, Tokyo
  - Eisai Trial Site 1, Ube-Shi, Yamaguchi
  - Eisai Trial Site 18, Chiba
  - Eisai Trial Site 15, Fukuoka
  - Eisai Trial Site 20, Kagoshima
  - Eisai Trial Site 19, Kochi
  - Eisai Trial Site 12, Kyoto
  - Eisai Trial Site 21, Niigata
  - Eisai Trial Site 24, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.